CLINICAL TRIAL: NCT06500923
Title: Five Year Outcomes at Two Narrow-diameter Implants to Replace Congenital Missing Maxillary Lateral Incisors
Brief Title: Narrow-diameter Implants Replacing Maxillary Lateral Incisors
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-58-0004
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ø2.9mm (Test): Test patients have received a 2.9 Ø dental implant
  Interventions: Other: Oral rehabilitation by means of implant-supported single unit crowns
- Ø3.3mm (Control): Control patients have received a 3.3 Ø dental implant
  Interventions: Other: Oral rehabilitation by means of implant-supported single unit crowns

INTERVENTIONS:
Other: Oral rehabilitation by means of implant-supported single unit crowns — Surgery: Implant placement; Prothetic rehabilitation: single unit crown

SUMMARY:
To present the 5-year clinical, radiographic, and aesthetic outcomes in patients with congenitally missing lateral incisors (MLIs) rehabilitated with two narrow-diameter implants (NDIs).

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by congenital missing with uni- or bilateral maxillary lateral incisors (i.e. 12 and/or 22)
* Patients with systemic health or controlled medical conditions
* Patients arrested skeletal growth as documented by two body height measurements at least one year apart not indicating continuous growth (Jensen, 2019)
* Written Informed Consent

Exclusion Criteria:

* Patients contraindications to implant therapy (Hwang & Wang, 2006, 2007) including
* Heavy smoking: >20 cigarettes/day
* Poor oral hygiene
* Compromised compliance
* Periodontally compromised conditions
* Patients with MLI's with the canine situated in the MLI region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by congenital missing with uni- or bilateral maxillary lateral incisors (i.e. 12 and/or 22)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Peri-implant marginal bone level changes | 1 year
  Changes in mm at the 1-year follow-up visit

SECONDARY OUTCOMES:
Implant Survival rate (%) | 1-3-5 year
  Number of implants in situ over the number of placed implants
Aesthetic outcomes | 1-3-5 year
  Evaluation of the aesthetic outcomes by means of a dedicated Index (Copenhagen Index Score CPI) (Score 1-4 / Score 1: best outcome; 4 : worst outcome)
PROMs | 1-3-5 year
  OHIP - 49 Scale (Score 1-3) (Score 1: best outcome; 3 : worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Storgaard Jensen, Prof., Study Chair — Copenhagen University Hospital, Copenhagen, Denmark
Locations (1):
- University Hospital Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No